CLINICAL TRIAL: NCT06856408
Title: Power of Growth RCT Study
Brief Title: Power of Growth - Digitally Assisted Intervention for the Early Childhood Educators' Self-efficacy Teamwork and Children's Behavioral Challenges.
Acronym: FinnPoG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Andre Sourander, MD Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PoG-001
Record Dates: First submitted 2025-02-13; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: ECE Teachers Self Efficacy; Team Work; Positive Pedagogy; Behavior Problems
Keywords: ECE self efficacy; team work; positive pedagogy; behavior problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digitally assisted intervention including online coaching (Experimental): The intervention is a structured remote coaching concept for professionals working in early childhood education. The intervention will use virtual reality glasses and 360° video material. The intervention consists of six self-study themes about positive pedagogy and team work. The themes will be combined with remote coaching for the team (3-5 people) and the skills will be practiced with their own group of children. The intervention length is 2-3 months. There will approximately 34 teams in intervention and control groups.
  Interventions: Behavioral: FinnPog
- Control (No Intervention): No digital assisted intervention or online coaching.

INTERVENTIONS:
Behavioral: FinnPog — The aim of the study is to find out how intervention affects the early childhood educators' self-efficacy teamwork and the changes in children's behavioral challenges. This RCT study has two parallel groups where teams of the daycare centres are randomized to intervention or control group. The research data is collected using electronic surveys and interviews.
  Arms: Digitally assisted intervention including online coaching

SUMMARY:
This is an RCT study investigating the efficacy of digital intervention focusing on enhancing positive directing skills for teams of early childhood education (ECE) professionals. The aims are to study 1) changes in the ECEs' self-assessed self-efficacy experience in the intervention group compared to the control group; 2) changes in the behavioral challenges of the children in the ECEs' groups assessed by the parents in the intervention group compared to the control group; and 3) changes in the ECEs' guidance methods in the intervention group compared to the control group. We will also study changes in the wellbeing of ECEs and teamwork in both treatment groups. The sample size will consist of approximately 64 teams of ECEs. Hence, altogether there will be approximately 200 study subjects.

The intervention is aimed at ECE teams and its goal is to strengthen and unify the team positive guidance practices in children's groups. The intervention includes self-learning material and teams online coaching in which the entire team participates simultaneously. The self-material includes 360 videos of everyday situations in the daycare and videos can be watched with VR glasses. The participants practice the skills systematically with their group of children. The duration of the intervention is approximately 12 weeks and team coaching are carried out approximately every two weeks.

ELIGIBILITY:
Inclusion Criteria:

Participant is working in a daycare centre team that is participating to the study. Sufficient knowledge in Finnish language.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
ECE Teacher Self Efficacy | From baseline to 3, 6 months after randomisation
  TEIP (Teacher Efficacy for Inclusive Practices)

SECONDARY OUTCOMES:
Perceptions of Team work | From baseline to 3, 6 months after randomisation
  TeamSTEPPS
Behaviour problems of the child | From baseline to 3, 6 months after randomisation
  Parent evaluates (SDQ, ARI, ICU)
Burn out | From baseline to 3, 6 months after randomisation
  BBI -15 (Bergen burnout inventory)
Confidence in ability to deal with child´s challenging behavior | From baseline to 3, 6 months after randomisation
  Questions about professional´s perceived confidence in ability to deal with child´s challenging behavior
Work satisfaction | From baseline to 3, 6 months after randomisation
  Questions about perceived work satisfaction
Perceived skills | From baseline to 3, 6 months after randomisation
  Questions about the content and themes of the intervention
Questionnaire on interaction skills: attuned interaction and guidance | From baseline to 3, 6 months after randomisation
  Questions about interaction skills
The workload of guiding the child group | From baseline to 3, 6 months after randomisation
  Questions about professional´s perceived workload of guiding the child group.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Early Childhood Education, Municipalities, Select
  - Research Centre of Child Psychiatry, Turku, Select